CLINICAL TRIAL: NCT07089316
Title: Preoperative MRI and Radiographic Parameters Are Associated With Medial Meniscus Posterior Root Tears and Predict Mid-Term Clinical and Radiographic Outcomes After Repair
Brief Title: Preoperative MRI and Radiographic Parameters in Medial Meniscus Root Tears and Repair Outcomes
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Fevzi Gurkan Aslan, Orthopaedic Surgery Resident, Department of Orthopaedics and Traumatology, Karadeniz Technical University Faculty of Medicine, Karadeniz Technical University
Other Study IDs: 24237859467
Record Dates: First submitted 2025-07-06; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Tibial Meniscus Tears
Keywords: Menisci, Tibial; Arthroscopy; Magnetic Resonance Imaging
MeSH Terms: conditions — Tibial Meniscus Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMPRT Patients: Patients with medial meniscus posterior root tears undergoing arthroscopic repair.
- Control Patients: Patients without meniscus tears, matched by age, BMI, and mechanical axis.

SUMMARY:
This retrospective observational study aims to investigate whether specific preoperative magnetic resonance imaging (MRI) and radiographic parameters are associated with medial meniscus posterior root tears (MMPRT), and whether these parameters have predictive value for mid-term clinical and radiographic outcomes after arthroscopic repair.

Patients with arthroscopically confirmed MMPRT treated between 2020 and 2024 are evaluated based on their preoperative MRI and standing knee radiographs. Imaging parameters of interest include medial tibial slope, meniscal extrusion, tibial plateau depth, posterior root angle, and intercondylar notch morphology. Clinical outcomes are assessed using standardized scoring systems. The study aims to identify imaging-based anatomical risk factors to improve diagnosis, patient selection, and prognosis following MMPRT repair.

DETAILED DESCRIPTION:
This retrospective observational study investigates the role of specific preoperative MRI and radiographic parameters in the diagnosis and prognosis of medial meniscus posterior root tears (MMPRT). Conducted at the Department of Orthopaedics and Traumatology, Karadeniz Technical University Farabi Hospital, the study aims to clarify whether morphologic imaging findings-such as medial tibial slope, meniscal extrusion, tibial plateau depth, posterior root angle, and intercondylar notch morphology-are associated with the presence of MMPRT and influence postoperative outcomes following arthroscopic repair.

All imaging measurements were performed using standardized techniques on MRI and radiographs obtained prior to surgery. Parameters were assessed by two independent orthopedic surgeons on separate occasions to evaluate interobserver reliability. A matched control group of patients without meniscal pathology was formed to strengthen the comparative analysis and support the identification of risk factors.

By analyzing a wide range of anatomic features on imaging, this study seeks to enhance early diagnostic accuracy, improve patient selection for surgical repair, and refine prognostic counseling. The findings are expected to contribute to the development of objective, imaging-based indicators that can guide clinical decision-making and predict mid-term clinical and radiographic outcomes after MMPRT repair.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older

Arthroscopically confirmed medial meniscus posterior root tear (MMPRT) diagnosis

Availability of preoperative knee MRI and standing long-leg radiographs

Minimum 24-month clinical and radiographic follow-up

Exclusion Criteria:

Lateral meniscus tear

Kellgren-Lawrence grade 3 or higher knee osteoarthritis

Advanced ligament injuries

History of previous knee surgery, osteotomy, or arthroplasty

Poor imaging quality

Mechanical axis deformities (varus or valgus alignment)

Follow-up period less than 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients diagnosed with medial meniscus posterior root tear (MMPRT) who underwent arthroscopic repair at Karadeniz Technical University Farabi Hospital between 2020 and 2024, as well as control patients without meniscus tears who had knee MRI and standing radiographs available in the same period. Controls were matched to the MMPRT group based on age, BMI, and mechanical axis distribution to minimize confounding.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Medial Tibial Slope | Preoperative MRI assessment
  Measured in degrees (°) on sagittal MRI. It is the angle between the tangent to the medial tibial plateau and the anatomical axis of the proximal tibia, drawn using a line connecting the anterior and posterior cortices of the plateau.
Medial Meniscus Extrusion | Preoperative MRI assessment
  Measured in millimeters (mm) on coronal MRI. Defined as the distance from the outer margin of the medial meniscus to the edge of the tibial plateau
Tibial Plateau Depth | Preoperative MRI assessment
  Measured in millimeters (mm) on sagittal MRI. It is the perpendicular depth from the deepest point of the medial tibial plateau concavity to a reference line connecting the anterior and posterior cortical rims.
Intercondylar Notch Width | Preoperative MRI assessment
  Measured in millimeters (mm) on axial MRI images. Width of the intercondylar notch at the level of the popliteal groove.
Intercondylar Distance | Preoperative MRI assessment
  Measured in millimeters (mm) on axial MRI. The distance between the outer surfaces of the medial and lateral femoral condyles at the level of the intercondylar notch.
Medial Femoral Condyle Angle | Preoperative MRI assessment
  Measured in degrees (°) on sagittal MRI. It is the angle between the femoral anatomical axis and the curvature of the medial femoral condyle.
Notch Width Index (ICNW/ICD Ratio) | Preoperative MRI assessment
  A unitless ratio obtained by dividing the intercondylar notch width by the intercondylar distance on axial MRI at the level of the popliteal groove.
Notch Shape | Preoperative MRI assessment
  Morphological classification based on axial MRI. The intercondylar notch is categorized into A-type, U-type, or W-type based on its geometric configuration.
Presence of Osteophyte (Spur) | Preoperative MRI assessment
  Binary variable (Yes/No) indicating the presence of an osteophyte at the intercondylar notch on axial or sagittal MRI.
Medial Femoral Condyle Width (MFCW) | Preoperative MRI assessment
  Measured in millimeters (mm) on coronal MRI. The width of the medial tibial plateau at its maximum span.
Medial Tibial Plateau Width (MTPW) | Preoperative MRI assessment
  Measured in millimeters (mm) on coronal MRI. The width of the medial tibial plateau at its maximum span.
MFCW/MTPW Ratio | Preoperative MRI assessment
  Unitless ratio calculated by dividing medial femoral condyle width (MFCW) by medial tibial plateau width (MTPW) on coronal MRI.
Medial Femoral Condyle Distal Offset Distance | Preoperative MRI
  Measured in millimeters (mm) on sagittal MRI at the level of the medial femoral condyle midpoint (defined on coronal MRI) as the perpendicular distance from the intercondylar axis to the most distal point of the condyle.
Medial Femoral Condyle Posterior Offset Distance | Preoperative MRI
  Measured in millimeters (mm) on the same sagittal MRI slice as the distal offset, defined as the distance from the intercondylar axis to the most posterior point of the condyle.
MFC Distal / Posterior Offset Ratio | Preoperative MRI
  A unitless ratio calculated by dividing the medial femoral condyle distal offset distance by its posterior offset distance on sagittal MRI.

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Score | Preoperative and minimum 24-month postoperative follow-up
  Scored from 0 to 100, this subjective assessment evaluates knee symptoms, function, and ability to engage in sports activities. Higher scores indicate better outcomes.
Lysholm Knee Score | Preoperative and minimum 24-month postoperative follow-up
  Scored from 0 to 100, this questionnaire evaluates limping, support, locking, pain, swelling, stair climbing, and squatting. Higher scores indicate better knee function.
Tegner Activity Scale | Preoperative and minimum 24-month postoperative follow-up
  Activity level is rated on a scale from 0 (disability) to 10 (elite sports). Assesses the return to daily or sports-related physical activity.
Kellgren-Lawrence Grade Progression | Preoperative and minimum 24-month postoperative radiographs
  Graded on a 0-4 scale, this radiographic classification evaluates the severity of osteoarthritis. Progression indicates worsening joint degeneration.
Medial Joint Space Width (JSW) | Preoperative and minimum 24-month postoperative radiographs
  Measured in millimeters (mm) on standing AP radiographs as the minimum vertical distance between the medial femoral condyle and tibial plateau. Reflects cartilage loss or joint space narrowing.

CONTACTS AND LOCATIONS:
Overall Officials: Fevzi Gurkan Aslan, M.D., Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Orthopedic and Traumatology Department, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared for this study. Only aggregate results and statistical analyses will be published to protect patient confidentiality.